CLINICAL TRIAL: NCT03010033
Title: Effects of Pulmonary Rehabilitation and Airway Management on Short-term and Long-term Perioperative Results of Lobectomy in Smoker Patients With Lung Cancer
Brief Title: Effect of Pulmonary Rehabilitation on Perioperative Outcomes in Smoker Patients With Lung Cancer
Acronym: PREPOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RTS-001
Record Dates: First submitted 2016-12-26; First posted 2017-01-04 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Neoplasm
Keywords: pulmonary rehabilitation; lobectomy; smoker
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular care (No Intervention): [Control group] preoperative treatment: smoking cession, aerosol inhalation for expectorant and antiasthmatic, anti-infection therapy if necessary and regular rehabilitation-propaganda; postoperative treatment: regular postoperative treatment (anti-infection, pain control, oxygen Inhalation aerosol inhalation for expectorant and antiasthmatic), patting back (3 times/day, 15min/time) and early ambulation unless serious patients.
- pulmonary rehabilitation (Experimental): [Study group] preoperative treatment: smoking cession, aerosol inhalation for expectorant and antiasthmatic, anti-infection therapy if necessary, regular rehabilitation-propaganda and interventional pulmonary rehabilitation (preoperative part); postoperative treatment: regular postoperative treatment (anti-infection, pain control, oxygen Inhalation aerosol inhalation for expectorant and antiasthmatic), patting back (3 times/day, 15min/time), early ambulation unless serious patients and interventional pulmonary rehabilitation (postoperative part).
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — pulmonary rehabilitation (preoperative part): lower extremity endurance training (using bike ergometer for 3 days, 2 times/day, 15-20min/time) or stair climbing training (3 days, 2 times/day, 30min/time), keep dyspnea index (Borg) score between 5 to 7 points. And inspiratory muscle training (using threshold inspiratory muscle trainer for 3 days, 5 times/day, 2 sessions/time, every session includes 10-20 cycle respirations).
  pulmonary rehabilitation (postoperative part): inspiratory muscle training (using threshold inspiratory muscle trainer until hospital discharge, 3-5 times/day, 1 session/time, every session includes 10-20 cycle respirations).
  Arms: pulmonary rehabilitation

SUMMARY:
It is reported that smoker patients (>400 cigarette/year) will suffer more postoperative complications than non-smoker patients after lobectomy. Evidences has suggested pulmonary rehabilitation could reduce the pulmonary complications after thoracic surgery. However, the effect and long-term results of pulmonary rehabilitation on smoker patients have not been studied. The purpose of this study is to determine whether pulmonary rehabilitation is effective to smoker patients who underwent lobectomy.

DETAILED DESCRIPTION:
In China, the smoker population is about 300 hundred million. Tobacco has become one of the world's public health problem. 30 percent of global surgery patients have smoking history. It is reported that smoker patients (>400 cigarette/year) will suffer more postoperative complications than non-smoker patients after lobectomy (38.2% vs 12.5%). Smoking is an independent risk factor of postoperative complications of cardiothoracic surgery. Evidences showed that smoking had a negative effect on airway management which plays an important role in postoperative recovery for thoracic surgery. Therefore, we hypothesise that intervention-related study to find a way to reduce postoperative complications for smoker patients is significantly meaningful in improving the overall outcome after pulmonary surgery as 80 percent of patients with lung cancer are smoker in China. Recently, a series of strategies on airway management have been proposed by clinical doctors. As one of the important parts of airway management, pulmonary rehabilitation has been demonstrated by evidence-base medicine to reduce the pulmonary complications after thoracic surgery and increase the breathing capacity. According to the reported literatures, the effect and long-term results of pulmonary rehabilitation on smoker patients have not been studied, so we designed this randomized controlled trial to determine whether pulmonary rehabilitation would be effective to smoker patients who underwent lobectomy which was associated with significant loss of lung function.

According to the reported papers in China, main observation index in experimental group was about 25.7, and in control group was about 10%. At the level of α=0.05 (Bilateral), power of test (1-β)=0.80, ratio=1:1. The estimated minimum required sample size of each group was 93 cases, the statistical loss rate was set as 10%. The overall sample size of this study was about 200 cases.

ELIGIBILITY:
Inclusion Criteria:

1. signed consent
2. smoker, ≥400/cigarette year
3. surgical approach: open or Video-assisted Thoracoscopic Surgery (VATS) lobectomy

Exclusion Criteria:

1. Serious physical diseases in patients during hospitalization, such as severe heart and lung diseases (CLASS III-IV) (FEV1/FVC <0.7and FEV1 <50% predicted value), kidney disease (ESRD change need to continue dialysis), or liver diseases (cirrhosis of the liver accompanied by ascites)
2. unable to obey interventional instructions/treatments because of any reasons
3. stage IV lung cancer
4. emergency surgery
5. lung cancer with preoperative chemotherapy, radiotherapy or chemoradiotherapy

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | postoperative in-hospital stay up to 30 days

SECONDARY OUTCOMES:
length of stay (LOS) | postoperative in-hospital stay up to 90 days
therapeutic time of antibiotics | Postoperative in-hospital stay up to 30 days
arterial blood gas analysis | before treatment, 3 days after treatment, 1 day after surgery, 3 days after surgery
vital signs | before treatment, 3 days after treatment, 1 day after surgery, 3 days after surgery
pain score of expectoration | 1 day and 3 days after surgery
  Visual Analogue Scale (VAS) Pain Score
amount of expectoration drainage | postoperative in-hospital stay up to 30 days
peak expiratory flow | before treatment, 3 days after treatment, 1 day after surgery, 3 days after surgery
lung function test | before treatment, 3 days after surgery, 3 months after surgery, 6 months after surgery
total hospitalization expenditures | postoperative in-hospital stay up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: He-Cheng Li, doctor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Han D, Wang X, Sun X, Cao Y, Li C, Guo W, Hu Y, Hang J, Li J, Xie Q, Li H. Ultra-short-period perioperative pulmonary rehabilitation on short-term outcomes after surgery in smoking patients with lung cancer: a randomized clinical trial. Int J Surg. 2025 Jan 1;111(1):581-588. doi: 10.1097/JS9.0000000000001856. PMID 38905498